CLINICAL TRIAL: NCT00770536
Title: A Phase 1b Study of AMG 386 in Combination With Either Pegylated Liposomal Doxorubicin or Topotecan in Subjects With Advanced Recurrent Epithelial Ovarian Cancer
Brief Title: AMG386 Comb w. Either Pegylated Liposomal Doxorubicin or Topotecan Subjects w. Advanced Recurrent Epithelial Ovarian CR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070182
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Cancer; Carcinoma; Fallopian Tube Cancer; Gynecological Malignancies; Metastases; Oncology; Ovarian Cancer; Solid Tumors; Tumors
Keywords: fallopian tube cancer; Gynecological Malignancy; primary peritoneal cancer of predominantly epithelial origin; Stage II to IV ovarian cancer
MeSH Terms: conditions — Neoplasms; Carcinoma; Fallopian Tube Neoplasms; Neoplasm Metastasis; Ovarian Neoplasms | interventions — liposomal doxorubicin; trebananib; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): In part 1, six subjects will be assigned to each cohort A or B. This is a dose escalation/de escalation study with a 6 + 3 design based on the incidence of DLTs (dose limiting toxicities) during the first 4 weeks of combined therapy [(cohort A: AMG 386 and pegylated liposomal doxorubicin) or (cohort B: AMG 386 and topotecan)].
  Interventions: Drug: A1: AMG 386 10 mg/kg + Liposomal doxorubicin; Drug: A3: AMG 386 15mg/kg + Liposomal doxorubicin; Drug: B1: AMG 386 10 mg/kg + Topotecan; Drug: B3: AMG 386 15mg/kg + Topotecan
- Part 2 (Experimental): The decision on declaration of a safe and tolerable dose during part 1 will lead to part 2 (cohort A: liposomal doxorubicin + AMG 386 MTD (max tolerated dose) of part 1, cohort B: Topotecan + AMG 386 MTD (max tolerated dose) of part 1
  Interventions: Drug: A1: AMG 386 10 mg/kg + Liposomal doxorubicin; Drug: A3: AMG 386 15mg/kg + Liposomal doxorubicin; Drug: B1: AMG 386 10 mg/kg + Topotecan; Drug: B3: AMG 386 15mg/kg + Topotecan

INTERVENTIONS:
Drug: A1: AMG 386 10 mg/kg + Liposomal doxorubicin — Liposomal doxorubicin 50 mg/m2 IV Q4W in combination with AMG 386 10 mg/kg IV QW
  Other Names: Liposomal doxorubicin; AMG 386
Drug: A3: AMG 386 15mg/kg + Liposomal doxorubicin — A3: AMG 386 15 mg/kg IV QW + Liposomal doxorubicin 50 mg/m2 IV Q4W
  Other Names: AMG 386; Liposomal doxorubicin
Drug: B1: AMG 386 10 mg/kg + Topotecan — B1: AMG 386 10 mg/kg IV QW + Topotecan 4 mg/m2 IV days 1, 8, 15, of a 28 day dosing schedule
  Other Names: Topotecan; AMG 386
Drug: B3: AMG 386 15mg/kg + Topotecan — AMG 386 15mg/kg IV QW + Topotecan 4mg/m2 IV days 1, 8, 15 of a 28 day dosing schedule
  Other Names: AMG 386; Topotecan

SUMMARY:
This study is a 2 part, 2 cohort, open-label, dose escalation/de escalation study of AMG 386 in combination with either pegylated liposomal doxorubicin or topotecan in subjects with recurrent ovarian cancer. Up to 100 subjects will be enrolled to receive AMG 386 in combination with either pegylated liposomal doxorubicin every 4 weeks (cohort A) or topotecan weekly on days 1, 8, and 15 of a 28 day dosing schedule (cohort B). Subject enrollment and assignment to either cohort will be based on eligibility and the investigator's discretion.

It is hypothesized that AMG 386, in combination with each of the chemotherapy regimens: either pegylated liposomal doxorubicin or topotecan will be safe and well tolerated in subjects with recurrent ovarian cancer.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness and safety of AMG 386 when used with pegylated liposomal doxorubicin or topotecan in subjects with advanced recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented recurrent invasive epithelial ovarian, fallopian tube, or primary peritoneal cancer
* Subjects must have received at least one platinum containing regimen
* Radiographically documented progression per RECIST criteria with modifications or progression of CA 125 as adopted by GCIG during or subsequent to the last chemotherapy regimen
* Subjects may include those with measurable or non measurable disease
* All scans and x-rays used to document measurable or non measurable disease must be done within 28 days prior to enrollment
* Female 18 years of age or older at the time the written informed consent is obtained
* GOG Performance Status of 0 or 1
* Left Ventricular Ejection Fraction (LVEF) >= institutional lower limit of normal for subjects assigned to cohort A only
* Adequate organ function as assessed by laboratory studies (hematological and chemistries)
* Life expectancy >= 3 months (per investigator opinion)
* Subjects of child bearing potential who have not undergone a bilateral salpingo oophorectomy and are sexually active must consent to use an accepted and effective double barrier non hormonal method of contraception from signing the informed consent through 6 months after last dose of study drug

Exclusion Criteria:

* Subjects believed to be a higher than average risk of bowel perforation. This includes symptoms of partial or complete bowel obstruction, recent (within 6 months) history of fistula or bowel perforation, subjects requiring total parenteral nutrition and continuous hydration
* Previous abdominal /or pelvic external beam radiotherapy
* Known history of central nervous system metastases
* Subjects with a history of prior malignancy, except:

  * Malignancy treated with curative intent and with no known active disease present for >= 3 years before study day 1 and felt to be at low risk for recurrence by treating physician
  * Adequately treated non melanomatous skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
* Prior myeloablative high dose chemotherapy with allogeneic or autologous stem cell (or bone marrow) transplant
* History of arterial or deep venous thromboembolism within 12 months prior to enrollment
* Clinically significant cardiac disease within 12 months prior to enrollment
* Prior treatment with doxorubicin or pegylated liposomal doxorubicin (cohort A subjects) and topotecan (cohort B subjects)
* Current or within 30 days prior to enrollment treatment with immune modulators such as systemic cyclosporine and tacrolimus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary objective is to identify the incidence of adverse events and clinical laboratory abnormalities defined as dose limiting toxicity in subjects treated with AMG 386 + pegylated liposomal doxorubicin (cohort A) and with AMG 386 + topotecan | first 4 weeks of treatment

SECONDARY OUTCOMES:
To evaluate the treatment effect as measured by: objective response rate (ORR), duration of response (DOR), PFS, change in tumor burden, CA 125 Response and Progression by GCIG and CA-125 duration of response | Treatment and follow-up phase of study
To evaluate the incidence of adverse events and clinical laboratory abnormalities not defined as DLTs. | first 4 weeks of treatment
To determine the pharmacokinetics of pegylated liposomal doxorubicin (and its metabolite, doxorubicinol), topotecan and AMG 386 (Cmax, AUC, and Cmin for intensive assessment; Cmax and Cmin for sparse assessment). | Treatment and follow-up phase of study
To estimate the incidence of anti AMG 386 antibody formation. | Treatment and follow-up phase of study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (16):
- United States (9):
  - Research Site, Tucson, Arizona
  - Research Site, Sacramento, California
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
- Australia (3):
  - Research Site, Adelaide, South Australia
  - Research Site, Footscray, Victoria
  - Research Site, Parkville, Victoria
- Belgium (4):
  - Research Site, Leuven
  - Research Site, LiÃ¨ge
  - Research Site, Liège
  - Research Site, Wilrijk

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com